CLINICAL TRIAL: NCT03578341
Title: Effect of Early Oral Colostrum Administration Versus Placebo on the Immune System in Premature Newborns Under 32 Weeks of Gestation: A Randomized Clinical Trial.
Brief Title: Oral Colostrum and Its Effect on Immune System
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Responsible Party: Principal Investigator, Silvia Romero-Maldonado, NEONATOLOGIST, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: 212250-2320-10305-01-16
Record Dates: First submitted 2018-06-22; First posted 2018-07-06 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Immune System Diseases; Premature Infant Disease; Immunoglobulin Deficiency
Keywords: Immunoglobulins A, G and M; Neonatal Sepsis; Human Milk; Orally Colostrum
MeSH Terms: conditions — Immune System Diseases; Agammaglobulinemia; Neonatal Sepsis

STUDY DESIGN:
Intervention Model Description: Intervention Model Description: The Participants will be randomly and assigned to Group 1, or Group 2 . using a table of random numbers, generated by a computer. The Human Milk Bank Staff, will prepares the colostrum and water (placebo) doses in syringes in such a way that it is not detected that it contains each of them, . Group 1: Will receive 0.3 mL orally colostrum every 4 h during three days, Group 2: will receive 0.3 mL orally Sterile water. Serum immunoglobulins A, G and M concentration will be determined before de start the orally doses, day 7 and 28 days of life.he nurse in charge of the patient's care, administer the dose, a doctor will take the laboratory exams and another researcher will collect and analyze the data. The syringes will be covered, to prevent the patiente´s nurse from observing the contents.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking Description: The colostrum and placebo will be preparing by a Human Milk Bank person, who will be knowing the treatment of both 2nd and 1st group. Both colostrum and placebo, will be administrating by nursing staff in syringes in such a way that it is not detected that it contains each of them. Neither the parents of the participants nor the researchers will be involved in the care or analysis of the data, until the end of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colostrum (Experimental): Group 1:(Colostrum): Preterm infants under 32 SDG will receive orally colostrum 0.3 mL every 4 h during three days.
  Interventions: Biological: Orally Colostrum
- Placebo (Placebo Comparator): Group 2: (Placebo): Preterm newborns under 32 SDG who will receive orally sterile water 0.3 mL every 4 h during three days.
  Interventions: Biological: Orally Colostrum

INTERVENTIONS:
Biological: Orally Colostrum — Group 1, Will receive colostrum 0.3 mL every 4 hours in the oropharyngeal mucosa, for 3 days.

SUMMARY:
The purpose of this project is to increase the serum immunological defenses of premature infants less then 32 weeks of gestation by administrating colostrum in the oropharyngeal mucosa versus placebo

DETAILED DESCRIPTION:
Prematurity is a public health problem because premature newborns have an immature immune system. Breast milk (colostrum) contains bioactive components that provide antimicrobial, anti-inflammatory, antioxidant, and immunomodulatory functions. These bioactive components are in higher concentrations in mothers' colostrum of premature babies. Because of the morbidities presented by premature infants, they remain fasting and lack the potential benefit provided by colostrum. When the colostrum is placed in the oropharyngeal mucosa, the immunocompetent cells stimulate the immune system, increasing the serum concentrations of immunoglobulins.

Objectives: To determine the efficacy of early administration of colostrum in the oropharyngeal mucosa in preterm infants less than 32 weeks of gestation and its effect on the immune system by quantifying immunoglobulins in preterm infants born at the National Institute of Perinatology. .

Methods / Design: 1 year, double blind randomized controlled clinical trial. The newborns included will be randomly assigned to one of the 2 groups: Group 1:, newborns receiving colostrum 0.3 mL every 4 hours in the oropharyngeal mucosa, for 3 days.

Newborns from Block B will receive orally sterile water (placebo) 0.3 mL following the same protocol. Serum immunoglobulin A, M and G concentrations will be determined before the start of the study on day 0 of life and after 7 and 28 days of life. They will continue in time until 36 SDG or at discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* NEWBORN 32 Gestational weeks
* Hospitalized in neonatal intensive care Unit
* Agreement signed by the legal representative

Exclusion Criteria:

* Intraventricular haemorrhage II/IV grade
* Congenital sepsis (early sepsis)
* Congenital malformations
* Early transfusions

Ages: 12 Hours to 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantification of serum Immunoglobulins | From baseline to day 7
  Quantification of immunoglobulins IgA, IgG and IgM

SECONDARY OUTCOMES:
sepsis neonatal | 28 days of postnatal age
  Frequency of neonatal sepsis
Necrotising Enterocolitis | 28 days of postnatal age
  Frequency of neonatal
Quantification of serum Immunoglobulins | From baseline to day 28
  Quantification of immunoglobulins IgA, IgG and IgM

CONTACTS AND LOCATIONS:
Overall Officials: Martha Morelos-Gonzalez, Chem, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes; Diana M Soriano-Becerril, MSc, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes; Jorge A Cardona-Pérez, MD, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes; Araceli Montoya-Estrada, PhD, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes; Elsa Castro-Millán, Thec, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes; Enrique Segura -Cervantes, MSc, Study Chair — Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Locations (2):
- Mexico (2):
  - Guadalupe del Carmen Estrada-Gutierrez, Miguel Hidalgo, Mexico City
  - Silvia Romero-Maldonado, Miguel Hidalgo, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Patients will be registered in a SPSS database
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The Data will be available in 2019, after the protocol is finished, for a month

REFERENCES:
- [Derived] Romero-Maldonado S, Soriano-Becerril DM, Garcia-May PK, Reyes-Munoz E, Munoz-Ortiz EG, Carrera-Muinos S, Granados-Cepeda ML, Cardona-Perez JA, Castro-Millan E, Segura-Cervantes E, Ceballos G, Montoya-Estrada A. Effect of Oropharyngeal Administration of Colostrum in Premature Newborns </=32 Weeks of Gestation on the Immune Response and Neonatal Morbidity: A Double-Blind Randomized Clinical Trial. Front Pediatr. 2022 Jul 8;10:891491. doi: 10.3389/fped.2022.891491. eCollection 2022. PMID 35874579